CLINICAL TRIAL: NCT06458504
Title: Virus-induced Immunosuppression Via Infection of Hematopoietic Progenitors
Brief Title: Viral Infection of HSPC Impacts Hematopoiesis
Acronym: MEGAHOST
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240419; 2024-A00117-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: HIV-1; SARS-CoV-2
Keywords: HIV-1; SARS-CoV-2; Hematopoietic Progenitors; Virus-induced; Immunosuppression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We propose to demonstrate that HIV-1 and SARS-CoV-2 are capable of targeting long-lived HSPC with self-renewal capacities. These progenitors, thus transformed into host cells, can give rise to a durable source of infected cells with an impact on hematopoiesis.

DETAILED DESCRIPTION:
Virus-induced immunosuppression is the transient or persistent decline of immune cell counts and/or function caused by a virus, favouring its persistence in the host organisms. When sustained, triggered by acute viral replication or maintained by chronic viral infections, virus-induced immunosuppression is a life-threatening condition. It is notoriously observed in chronic HIV-1 infection and even in a considerable fraction of antiretroviral-treated HIV-infected individuals. It is also observed in some individuals recovering from severe and mild-to-moderate COVID-19. Its mechanisms are elusive and efficient therapeutic options are not available. Virus-induced immunosuppression may occur in the periphery (affecting circulating immune cells) or in the bone marrow, affecting hematopoietic stem and progenitor cells (HSPC) and hematopoiesis. Several viruses can infect HSPCs. HIV-1 can directly infect HSC, negatively impacting HSC function and the whole stem cell environment of the bone marrow. Whether HSC can be productively infected by SARS-CoV-2 or just targeted and modulated by it remains uncertain and further studies are required to determine HSPC susceptibility or viral sensing for SARS-CoV-2. Therefore, we will i) Evaluate which hematopoietic stem and progenitor cells (HSPC) are targeted by HIV-1 (in vivo and ex vivo) and SARS-CoV-2 (ex vivo); ii) Evaluate whether these infected HSPC would modulate the bone marrow environment by upregulating inflammatory cytokines detrimental to lymphopoiesis.

ELIGIBILITY:
Inclusion Criteria:

HIV patients :

* HIV-positive patients with a negative or positive viral load.
* managed at Ambroise Paré Hospital.
* patients with a bone marrow biopsy or myelogram performed as part of their care.

Healthy subjects without HIV - patients with a BM biopsy or myelogram performed as part of their care for a suspected hematological pathology.

Management at Ambroise Paré Hospital.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * adult patients.
  * patients able to read and understand the information note.
  * no opposition to the use of biological samples. 45 subjects are required in our study:
  (A) 20 patients with FFPE osteomedullary biopsy prior to COVID-19 pandemic. Including :
  * 10 HIVpos patients selected based on biopsy results (normal, subnormal/minor lesion).
  * 10 HIVneg patients selected to match HIVpos patients, considering age and biological sex.
  (B) 25 HIVneg patients asymptomatic for COVID-19 for whom a myelogram or BM biopsy is prescribed as part of a search for haematological pathology or as part of lymphoma extension investigations.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate if infected HSPC would modulate the bone marrow environment | at 1 year
  Evaluate whether these infected HSPC would modulate the bone marrow environment by upregulating inflammatory cytokines detrimental to lymphopoiesis.

CONTACTS AND LOCATIONS:
Overall Officials: Claude CAPRON, MD, PhD, Principal Investigator — Laboratory of Immunology, Ambroise Paré hospital - APHP; Fernando REAL, PhD, Study Director — Center for Infection and Immunity of Lille, INSERM U1019 - CNRS UMR9017, Institut Pasteur de Lille
Locations (1):
- Hematology and interne medicine department, Ambroise Paré hospital - APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: Undecided